CLINICAL TRIAL: NCT00601068
Title: Proposal For The Development Of A Well Defined Database For Patients With Oral Bisphosphonate-Related Osteonecrosis of the Jaws (BON)
Brief Title: Proposal For The Development Of A Well Defined Database For Patients With Oral Bisphosphonate-Related Osteonecrosis
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 32936; 00065255 UFID
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2012-07

CONDITIONS: Osteonecrosis
Keywords: osteonecrosis, jaws, bisphosphonate, fosamax, alendronate
MeSH Terms: conditions — Osteonecrosis | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — biopsy tissue submitted from bone biopsies
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational: Group of patients with osteochemonecrosis related to oral bisphosphonate use
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Group of patients with osteochemonecrosis related to oral bisphosphonate use
  Other Names: Osteochemonecrosis

SUMMARY:
In cooperation with Merck & Co, Inc. we will identify and form a database of 35 patients who have developed osteochemonecrosis of the jaws related to oral bisphosphonate use. We will study the triggers, associated medical conditions and medications, location of the lesion(s), and patient outcomes.

DETAILED DESCRIPTION:
This study is an observational study, and not a comparative trial. The major outcome is represented by the fraction of subjects with long term healed lesions.

ELIGIBILITY:
Inclusion Criteria:

* Exposed bone in the oral cavity of greater than 6-8 weeks duration unresponsive to therapy

Exclusion Criteria:

* Pregnant patients
* Patients less than 30 yrs of age or greater than 90 yrs of age
* Mentally incompetent individuals

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who develop exposed bone in their mouth and are on an oral bisphosphonate
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2007-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
establish complete database and publish descriptive paper | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Donald M Cohen, DMD, MS, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States